CLINICAL TRIAL: NCT01615549
Title: Proficiency-based Versus Free Laparoscopic Training in Cholecystectomy Using the Simbionix LAP Mentor™. A Randomized Controlled Trial
Brief Title: Efficacy of Proficiency-based Versus Free Laparoscopic Training in Cholecystectomy on a Virtual Reality Simulator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Bonn (Other); University Hospital, Basel, Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Simbionix 20120507; SNSF 32003B-120722 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF))
Record Dates: First submitted 2012-05-23; First posted 2012-06-08 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Cholelithiasis; Cholecystitis; Cholecystolithiasis
Keywords: Cholecystectomy; Virtual reality device; Training
MeSH Terms: conditions — Cholelithiasis; Cholecystitis; Cholecystolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Free training (Active Comparator)
  Interventions: Procedure: Laparsocopic cholecystectomy
- Proficiency-based training (Experimental)
  Interventions: Procedure: Laparsocopic cholecystectomy

INTERVENTIONS:
Procedure: Laparsocopic cholecystectomy — Perform laparsocopic cholecystectomy on a virtual reality devise
  Other Names: Key whole gall bladder surgery

SUMMARY:
Virtual reality devices are widely accepted tools to familiarize surgical novices with the principles of laparoscopy. Free Virtual reality training will be tested against basic training and efficacy assessed in a randomized controlled trial of surgical novices.

DETAILED DESCRIPTION:
Virtual reality simulators are widely accepted tools to familiarize surgical novices with the principles of laparoscopy without jeopardizing patient safety. However, access to a Virtual reality simulator and initial instruction alone followed by free training of the surgical novice may not be sufficient to achieve the training goals efficiently. The aims of this study are to determine if proficiency based laparoscopic training on the Simbionx LAP Mentor™ with external formative assessment using peer group derived benchmarks is superior to free training with self-assessment using the simulated laparoscopic cholecystectomy procedure with different endpoints (time to extract the gallbladder, serious complications, safe cautery and instrument pathways) as outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Surgical novices (trainees / residents)
* Performed less than five laparoscopic procedures
* No previous simulator experience

Exclusion Criteria:

* Specialist surgeons
* Performed more than five laparoscopic procedures
* Previous experience with a simulator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2004-04; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to extract the gall bladder. | 10 minutes in average
  The time to extract the gall bladder on a virtual simulator is typically 10 minutes. However this varies according to the settings of the difficulty chosen on the virtual reality software. This is a continuous variable measuring the duration for a trainee surgeon to extract the gall bladder (measured in seconds). The start point is the beginning of the exercise and the finishing point is once the gall bladder is completely resected (gall bladder mobilized and the cystic duct and artery dissected and ligated).

SECONDARY OUTCOMES:
Serious intra-operative complications | 10 minutes in average
  Serious complications on a virtual simulator are considered injuries to the bile duct, hepatic artery, the bowel, or the liver bed. Such complications are automatically detected by the virtual reality software and recorded in a special database. This is a continuous variable with "0" indicating no complications, "1" indicating one complication, "2" indicating two complications, etc.
Safe cautery | 10 minutes in average
  During a virtual laparoscopic cholecycetoctomy, cautery (also know as a coagulator, a device that utilizes electrical current for dissection or bleeding control)is commonly used to mobilize the gall bladder away from the liver bed. The virtual simulator software measures the percentage of the unsafe use of cautery. This is a continuous variable with 100% safe cautery indicating no unsafe cauterization around important structures such as the bowel, bile duct, hepatic artery, etc.
Total path length of right instrument | 10 minutes in average
  The total path length of the right instrument used to extract the gall bladder during a virtual laparoscopic cholecystectomy task measures the "in and out" movement of the right instrument. The higher the value, the more unnecessary movements are made during the task.

CONTACTS AND LOCATIONS:
Overall Officials: Martin W von Websky, MD, Principal Investigator — University Hospital Zurich, Department of Surgery; Dimitri A Raptis, MD, MSc, Principal Investigator — University Hospital Zurich, Department of Surgery; Pierre-Alain Clavien, MD, PhD, Study Chair — University Hospital, Zürich; Dieter Hahnloser, MD, Study Director — University Hospital Zurich, Department of Surgery
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Zurich, Canton of Zurich
  - University Hospital Zurich, Department of Surgery, Zurich

REFERENCES:
- [Derived] von Websky MW, Raptis DA, Vitz M, Rosenthal R, Clavien PA, Hahnloser D. Access to a simulator is not enough: the benefits of virtual reality training based on peer-group-derived benchmarks--a randomized controlled trial. World J Surg. 2013 Nov;37(11):2534-41. doi: 10.1007/s00268-013-2175-6. PMID 23942532